CLINICAL TRIAL: NCT01222156
Title: Remote Intracardiac Catheter Target Acquisition Using the Magnetecs Catheter Guidance Control and Imaging (CGCI) System
Brief Title: Accuracy and Safety Study of the Magnetecs CGCI System for Intracardiac Mapping
Acronym: RICTAM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Magnetecs Corporation (Other)
Responsible Party: Josh Sachar/CEO and Chief Technology Officer, Magnetecs, Corp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CGCI HS01
Record Dates: First submitted 2010-10-14; First posted 2010-10-18 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-10

CONDITIONS: Tachycardia, Supraventricular; Tachycardia, Ventricular
Keywords: Cardiac arrhythmias; Catheter ablation; Electrophysiology; Magnetic; Mapping; Remote navigation
MeSH Terms: conditions — Tachycardia, Supraventricular; Tachycardia, Ventricular; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CGCI navigation (Experimental): Subjects with CGCI navigation to specific target intracardiac anatomical sites
  Interventions: Procedure: Remote magnetic navigation; Device: Magnetecs Catheter Guidance Control and Imaging system

INTERVENTIONS:
Procedure: Remote magnetic navigation — Remote magnetic navigation of electrophysiology catheters to target intracardiac anatomical sites at mapping-ablation procedures in patients with cardiac arrhythmias
  Other Names: Magnetecs; CGCI
Device: Magnetecs Catheter Guidance Control and Imaging system — Magnetecs Catheter Guidance Control and Imaging (CGCI) system

SUMMARY:
The Magnetecs Catheter Guidance Control and Imaging (CGCI) system is a magnetic remote navigation system which is comprised of a magnetic chamber of eight electromagnets around the patient torso. The system can change the magnetic field almost instantaneously and enables almost real time manipulation of a special magnetic catheter (Maxwell mapping catheter) which results in accurate, repeatable, rapid and safe target acquisition within the four chambers of the human heart.

The trial is a prospective, non-randomized, clinical one designed to test the study hypotheses of (a) technical equivalence of the study device in comparison to other magnetic remote navigation systems, (b) performance equivalence or non-inferiority of the study device target acquisition capability compared to presently used catheter navigation techniques, and (c) safety equivalence or non-inferiority of the study device in comparison to catheter navigation devices using other navigation techniques.

DETAILED DESCRIPTION:
The CGCI system is comprised of (a) magnetic chamber of eight electromagnets around the patient torso, (b) the Maxwell ©, a 7Fr. Inquiry™ catheter with an attached magnetic pellet manufactured by St. Jude Medical, Inc. The Maxwell © is equivalent to a 7 Fr. Inquiry™ cleared under 510(K) K022380, and (c) a Agilis ES Active Sheath© which is a modified 7.5 Fr. Steerable Introducer is equivalent to the Agilis NxT™ Steerable Introducer, manufactured by St. Jude Medical, Inc. and cleared under 510(K) K061363.

Study Rationale: Current manual manipulations of mapping catheters are imprecise and difficult to control. The Magnetecs CGCI system enables almost real time manipulation of the Maxwell mapping catheter which results in accurate, repeatable, rapid and safe target acquisition. The CGCI System is intended to navigate a magnetic catheter within the four chambers of the human heart by orienting and moving the catheter tip to designated anatomically significant targets.

Design: A prospective, non-randomized, clinical trial designed to test the study hypotheses of (a) technical equivalence of the study device in comparison to other magnetic remote navigation systems, (b) performance equivalence or non-inferiority of the study device target acquisition capability compared to presently used catheter navigation techniques, and (c) safety equivalence or non-inferiority of the study device in comparison to catheter navigation devices using other navigation techniques.

Target Population:Patients who have recurrent cardiac rhythm disturbances and who meet clinically recognized indications for performance of an intracardiac mapping procedure.

Planned Number of Subjects: A total of 40 patients

Study Objectives: This study is designed to collect data to test the target acquisition performance efficacy and safety of the CGCI for intracardiac navigation.

The objective is to achieve the navigation performance criteria for the primary efficacy endpoints for reaching preselected anatomically significant targets in the right and left heart chambers, respectively. The secondary efficacy endpoints are obtained by measurements of stimulation thresholds at selected anatomic sites, and by analyzing surface and intracardiac signal recordings during target acquisition with the CGCI magnetic system.

The primary safety endpoints are defined as the rate of procedure related incidence of serious acute Adverse Events due to manipulation of the magnetic catheter. Verification of these adverse events will be by fluoroscopy, echocardiograms and physician observations, and the results will be subjected to statistical evaluation.

The claims of substantial technical equivalence to other magnetic remote navigation systems will be verified by collecting data at the outset of each clinical procedure, measuring maximum magnetic field strength at the center region and around the outside perimeter of the CGCI device, and by measuring the maximum force available at the catheter tip.

Success will be evaluated in accordance with the primary efficacy and safety endpoint specifications, and by the technical equivalency tests. Data collection and sample size are defined to comply with FDA (1992) 80/20 ruling to adequately power the hypothesis tests.

Investigational Site: Hospital Universitario La Paz P. Castellana, 216. 28046 Madrid, Spain Tel/ Fax: + 34 917277564

Participating Physicians: Dr. Jose Luis Merino, Dr. Vivek Reddy, Dr. Eli Gang, Dr. Armando Perez Silva, Dr. Sara Moreno Reviriego, Dr. Sergio Castrejon, Dr. Alejandro Estrada, Dr. David Doiny, Dr. Bich-Lien Nguyen, Dr. Petr Neuzil, Dr. Andre D'Avila.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are clinically eligible for catheter based therapy of cardiac arrhythmias
2. Body Mass Index (BMI) < 40
3. Signed Informed Consent

Exclusion Criteria:

1. Indication for atrial fibrillation ablation
2. Indication for ischemic ventricular tachycardia ablation
3. Severe cerebrovascular disease
4. Serum creatinine >2.5
5. Active gastrointestinal bleeding
6. Active infection or fever
7. Short life expectancy (<6 months)
8. Severe uncontrolled systemic hypertension
9. Severe electrolyte imbalance
10. Congestive heart failure (NYHA Class IV)
11. Unstable angina
12. Recent MI (<4 weeks)
13. Bleeding or clotting disorders
14. Uncontrolled diabetes
15. Inability to receive IV Anticoagulants
16. Presence of intracardiac thrombus
17. Patients with prosthetic cardiac valves
18. Patients with permanent pacemakers or ICD's
19. Pregnancy
20. Enrollment in any other ongoing clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Intracardiac anatomic site target acquisition and repetition acquisition success rates | within 1 minute
  Intracardiac anatomic site target acquisition and repetition acquisition success rates of a mapping catheter remotely navigated by the Magnetecs CGCI system
Serious adverse event rate | within 7 days
  Serious adverse event rate at intracardiac anatomic site target acquisition of a mapping catheter remotely navigated by the Magnetecs CGCI system

SECONDARY OUTCOMES:
Intracardiac anatomic site target acquisition and repetition acquisition duration | within 1 minute
  Intracardiac anatomic site target acquisition and repetition acquisition duration of a mapping catheter remotely navigated by the Magnetecs CGCI system
Pacing stimulation thresholds levels at the target intracardiac anatomic sites remotely and manually acquired | within 10 minutes
  Pacing stimulation thresholds levels at the target intracardiac anatomic sites remotely and manually acquired by the Magnetecs CGCI system and a conventional catheter manually operated respectively.
Electrogram frequency spectrum and signal/noise levels at the target intracardiac anatomic sites remotely and manually acquired by the Magnetecs CGCI system and a conventional catheter manually operated respectively. | within 1 minute
  Electrogram frequency spectrum and signal/noise levels at the target intracardiac anatomic sites remotely and manually acquired by the Magnetecs CGCI system and a conventional catheter manually operated respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Merino, MD, PhD, Principal Investigator — Hospital Universitario La Paz; Eli Gang, MD, Study Director — Magnetecs, Corp; Vivek Y Reddy, MD, Study Chair — Mount Sinai Hospital, New York, USA
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

REFERENCES:
- See also: Sponsor website with information about the system and the trial — http://www.magnetecs.com